CLINICAL TRIAL: NCT02607501
Title: A Multi-center Post Marketing Study Evaluating the Safety, Technical Feasibility, and Efficacy of the eCLIPs™ Family of Products for the Treatment of Bifurcation Intracranial Aneurysms.
Brief Title: European eCLIPS™ Safety, Feasibility and Efficacy Study
Acronym: EESIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: Evasc Medical Systems Corp. (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-15-009
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Saccular Aneurysm; Intracranial Aneurysm
Keywords: coil embolization; bifurcation
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eCLIPs BRS (Other): Implant eCLIPs BRS at target aneurysm
  Interventions: Device: Implant eCLIPs

INTERVENTIONS:
Device: Implant eCLIPs — Implant eCLIPs at target bifurcation aneurysm

SUMMARY:
An open label, prospective, multicentre, single-arm, post marketing study evaluating the safety, technical feasibility, and efficacy of the eCLIPs™ Family of Products for the treatment of bifurcation intracranial aneurysms.

DETAILED DESCRIPTION:
The objective of this study is to obtain data on the technical feasibility, safety, and efficacy of the eCLIPs™ Products for the treatment of bifurcation aneurysms. Specifically, procedural success of the eCLIPs Bifurcation Remodelling System (BRS) will be evaluated to determine feasibility of this product and safety will be measured as of a major stroke or death within 30 days, or major territorial stroke or neurological death within one year. Additional endpoints will be evaluated and data collected to assess the procedural success of the other eCLIPs Products Microcatheter, Microintroducer, Detacher) and collect efficacy information on the eCLIPs Products. A rate of 69% of aneurysms achieving Raymond Class 1 occlusion at the 12 month endpoint has been chosen as the criterion for success in subjects treated with the eCLIPs Device and coils (primary endpoint).

An upper 95% confidence interval of 10% rate of major ipsilateral stroke or death at the 1 month, and 12 month endpoint has been chosen to demonstrate clinically safety (primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

1. Patient whose age is greater than 18 years old
2. Patient with an unruptured or previously ruptured (at least 1 month from date of rupture and with partial occlusion of the dome of the aneurysm by endovascular techniques or by open neurosurgery, and in stable neurological condition-WFNS I and II with a good recovery to at least to mRS 0-2) saccular, intracranial aneurysm or recurrent aneurysm, which arises at a bifurcation of Basilar Tip or Carotid Terminus and has a neck length of > 4mm or dome:neck ratio <2.
3. Patient aneurysm arises at a bifurcation artery with at least one of the two branch artery vessels having a diameter between 1.5mm and 3.25mm
4. Patient understands the nature of the procedure and has the capacity to provide informed consent.
5. Patient is willing to have on-site 30- day, 6-month, and 12 month follow-up evaluations as per standard clinical practice.

Exclusion Criteria:

1. Patient who presents with an intracranial mass or currently undergoing radiation therapy for carcinoma of the head or neck region.
2. Major surgery within previous 30 days or planned in the next 120 days after enrolment.
3. Patient with an International Normalized Ratio (INR)≥ 1.5.
4. Patient with serum creatinine level ≥104 µmol/L (or 2.5mg/dL) at time of enrolment.
5. Patient with a platelet count ˂100x103 cells/mm3 or known platelet dysfunction at time of enrolment
6. Patient who has a known cardiac disorder, likely to be associated with cardio-embolic symptoms such as atrial fibrillation
7. Patient with any condition that, in the opinion of the treating physician, would place the participant at a high risk of embolic stroke or with any medical co-morbidity likely to affect the outcome (e.g. pulmonary disease, uncontrolled diabetes, blood disorders).
8. Patient with known allergies to nickel-titanium metal
9. Patient with known allergies to aspirin, heparin, ticlopidine, clopidogrel, prasugrel or other anti-platelet or P2Y12 agents or to general anesthesia.
10. Subject has resistance to Prasugrel based on a validated platelet testing method (Verify Now, Multiplate or other).
11. Patient with a life threatening allergy to contrast (patients with itching or rash as a reaction to contrast can be included if properly prophylactically treated).
12. Patient with inappropriate anatomy as demonstrated by angiography due to severe intracranial vessel tortuosity or stenosis, or intracranial vasospasm not responsive to medical therapy.
13. Patient who is currently participating in another clinical research study involving an investigational product.
14. Patient who has had a previous intracranial procedure associated with the target aneurysm such that access and placement of an eCLIPS device would be compromised
15. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to the treatment date.
16. More than one intracranial aneurysm that requires treatment within 12 months.
17. Asymptomatic extradural aneurysms requiring treatment.
18. Severe neurological deficit that renders the subject incapable of living independently.
19. Unstable neurological deficit (i.e. worsening or improvement of clinical condition in the last 30 days.
20. Dementia or psychiatric problem that prevents the subject from completing required follow up.
21. Subject had a subarachnoid haemorrhage within 6 months prior to enrolment date.
22. Subject has a non-treated arterio-venous malformation in the territory of the target aneurysm.
23. Subject has a need for long-term use of anticoagulants.
24. Patient who is unable to complete the required follow-up.
25. Inability to understand the study or history of non-compliance with medical advice.
26. Evidence of active infection at the time of treatment.
27. Patient who is pregnant or breastfeeding.
28. Patient who has participated in a drug study within the last 30 days.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Safety End Point: absence of a major territorial stroke or death (procedural). | 30 days
  Major territorial stroke was defined as an ischemic or hemorrhagic stroke resulting in an increase of ≥4 points on the NIH Stroke Scale/Score (NIHSS) and that persisted for >24 hours.
  NIHSS ranges from 0 to 4; with lower scores indicating better outcome.
Absence of a major territorial stroke or neurological death | 31 days to 12 months
  Major territorial stroke was defined as an ischemic or hemorrhagic stroke resulting in an increase of ≥4 points on the NIH Stroke Scale/Score (NIHSS) and that persisted for >24 hours. NIHSS ranges from 0 to 4; with lower scores indicating better outcome.
Complete aneurysm occlusion (Raymond 1 ) | 6 months
  complete aneurysm occlusion (modified Raymond-Roy classification (mRRc) I), adjudicated by an independent core laboratory. mRRC ranges from 1 to 3b; where lower scores (1) indicate better outcome.
Complete aneurysm occlusion (Raymond 1 ) | 12 months
  complete aneurysm occlusion (modified Raymond-Roy classification (mRRc) I), adjudicated by an independent core laboratory. mRRC ranges from 1 to 3b; where lower scores (1) indicate better outcome.

SECONDARY OUTCOMES:
eCLIPs Bifurcation Remodeling System Technical Success | Procedural
  measured by the proportion of successful eCLIPs Device implants at the target aneurysm
Complete or near complete (Raymond 1 and 2) | 6 and 12 months
  complete aneurysm occlusion (modified Raymond-Roy classification (mRRc) I or II), adjudicated by an independent core laboratory. mRRC ranges from 1 to 3b; where lower scores (1) indicate better outcome.
Degree of Flow Diversion (reduction of blood flow into aneurysm) | immediately after eCLIPs implant, before coiling
  reduction of blood flow into aneurysm according to the O'Kelly-Marotta (OKM) grading scale
Success of adjuvant coiling into aneurysm after successful eCLIPs Device implant | Procedural
  Success of adjunctive coiling into aneurysm after successful eCLIPs implantation, assessed by the operator.
Change in Modified Rankin Score | from Baseline to 1 month, 6 months and 12 months
  Change in Modified Rankin Score (mRS) from baseline. The mRS ranges from 0 to 6; lower scores indicate better outcome.
Occurrence of unplanned aneurysm re-treatment | within 12 months
  endovascular or surgical repair
Assessment of Device Migration | at 6 months and 12 months
  Frequency of eCLIPs Device migration
Assessment of artery stenosis at the device location | at 6 months and 12 months
  Frequency of cases with artery stenosis at the device location
Assessment of artery patency at the target aneurysm | at 6 months and 12 months
  Frequency of cases with artery patency at the target aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Joost DeVries, M.D., Principal Investigator — Radboud University Medical Center
Locations (4):
- Aarhus Universitetshospital, Aarhus, Denmark
- Universitaetsklinikum Duesseldorf, Düsseldorf, Germany
- Netherlands (2):
  - Maastricht University Hospital, Maastricht
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Vries J, Aquarius R, Sorensen L, Boogaarts HD, Turowski B, van Zwam WH, Marotta TR, Bartels RHMA. Safety and efficacy of the eCLIPs bifurcation remodelling system for the treatment of wide necked bifurcation aneurysms: 1 year results from the European eCLIPs Safety, Feasibility, and Efficacy Study (EESIS). J Neurointerv Surg. 2023 Feb;15(2):163-171. doi: 10.1136/neurintsurg-2021-018460. Epub 2022 Apr 7. PMID 35393338